CLINICAL TRIAL: NCT00862381
Title: Opothérapie Par Hydrocortisone après Injection Unique d'Etomidate Chez le Patient de réanimation
Brief Title: Hydrocortisone Use After Etomidate in Intensive Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Dr Christophe BROUX, Pôle Anesthésie-Réanimation - CHU de Grenoble
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0726; 2007-007603-32 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Patient Admitted in Reanimation
Keywords: shock; Tracheal Intubation; reanimation; suprarenal insufficiency; Etomidate; Adrenocorticotropic Hormone; hydrocortisone
MeSH Terms: conditions — Shock | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Hydrocortisone
  Interventions: Drug: Hydrocortisone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — hemisuccinate d'hydrocortisone, 200mg per 24 hours, 48 hours of treatment
  Arms: 1
Drug: Placebo — NaCl 0.9%
  Arms: 2

SUMMARY:
the objective of the study is to assess the value of substitution with 200mg/24h of hydrocortisone for 48 hours for patients in intensive care who have received a single injection of etomidate

DETAILED DESCRIPTION:
Etomidate is a hypnotic widely used for patients in intensive care who require rapid induction, because of its short duration of action, its excellent cardiovascular tolerance and maintenance of cerebral perfusion pressure.

For this reason etomidate remains the hypnotic of choice for induction of unstable patients. Other hypnotics currently in existence do not provide adequate safety with a sufficiently predictable and stable effect in this situation. However, it may induce acute adrenal insufficiency by inhibition of 11-b-hydroxylase necessary for the synthesis of cortisol from compound S. An observational study conducted at the Grenoble University hospital in 2006 showed that the duration of this blockage can reach up to 48 hours. Acute adrenal insufficiency in intensive care patients is associated with a poor prognosis. The main objective of this study is to assess the value of substitution with 200mg/24h of hydrocortisone for 48 hours for patients in intensive care who have received a single injection of etomidate.

This is an interventional, prospective, randomized, placebo-controlled, double-blind, analytical study with a cohort of 100 patients between 18 and 80 years, of both sexes, who have had tracheal intubation in a pre-hospital or shock treatment setting with the administration of a single injection of etomidate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received an unique injection of etomidate in pre-hospital situation or at "déchocage" in the previous 6 hours.
* informed consent signed by the patient or the reliable person
* affiliation to a regime of social security

Exclusion Criteria:

* persons aimed at the articles L. 1121-5 à L. 1121-8 of the french code of public health
* toxic shock requiring a treatment by HSHC inn accordance with the criteria of Annane et Al. [13]
* purpura fulminans
* chronicle suprarenal insufficiency
* patients likely to present an acute suprarenal insufficiency : current treatment with antifungal : ketoconazole or fluconazole, known HIV infection, Sheehan syndrome
* corticotherapy in the 6 last months
* initiation of hydrocortisone therapy out of the study
* survival estimated at less than 48 hours
* no benefits of social security
* refusal to participate by patient or reliable person

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
diminution of 50% of the proportion of patients with a score SOFA of 3 or 4 | 12h, 24h and 48h after the injection of hydrocortisone
mean arterial blood pressure | during the hospitalisation
plasmatic cortisol and substance S before and after ACTH stimulation | h-4; h6; h12 and h24

SECONDARY OUTCOMES:
clinical state | 12h and 24h
hospitalisation duration in reanimation | until day28
duration of mechanical ventilation | until day28
duration and posology of adrenaline and noradrenaline | h0, h4, h6, h12, h24 and h48
complications during hospitalization in reanimation potentially due to HSHC | until day28
dose of etomidate injection | h0
mortality | day28

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PH, BROUX, Principal Investigator — University Hospital of Grenoble, France
Locations (2):
- France (2):
  - Réanimation polyvalente déchocage, centre hospitalier de la région Annecienne, Annecy
  - Pôle d'anesthésie - réanimation, University Hospital of Grenoble, Grenoble

REFERENCES:
- [Derived] Payen JF, Dupuis C, Trouve-Buisson T, Vinclair M, Broux C, Bouzat P, Genty C, Monneret D, Faure P, Chabre O, Bosson JL. Corticosteroid after etomidate in critically ill patients: a randomized controlled trial. Crit Care Med. 2012 Jan;40(1):29-35. doi: 10.1097/CCM.0b013e31822d7938. PMID 21926601